CLINICAL TRIAL: NCT07236801
Title: An Exploratory Clinical Study on the Safety and Efficacy of YTS109 Cell in Subjects With Relapsing/Refractory Autoimmune Diseases
Brief Title: Exploratory Clinical Study on YTS109 Cell Therapy for Autoimmune Diseases
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: China Immunotech (Beijing) Biotechnology Co., Ltd. (Industry)
Collaborators: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YTS109-009
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Systemic Lupus Erythematosus (SLE); Systemic Sclerosis; Sjogren's Syndrome (SS); Inflammatory Myopathy; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Antiphospholipid Syndrome
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Scleroderma, Systemic; Sjogren's Syndrome; Myositis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Antiphospholipid Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YTS109 cell (Experimental)
  Interventions: Drug: YTS109 cell

INTERVENTIONS:
Drug: YTS109 cell — Subjects will receive a single infusion of YTS109 cells. The dose groups are set to commence at 3×10⁶ STAR -T cells/kg, employing a 3+3 escalation principle for dose titration.

SUMMARY:
This study evaluates the safety and efficacy of YTS109 cells in adults with relapsed/refractory autoimmune diseases, such as Systemic Lupus Erythematosus (SLE), including LN and SLE-ITP, Sjogren's Syndrome, etc. Aproximately 18 patients aged 18-65 will receive a single infusion of YTS109 cells. The dose groups are set to commence at 3×10⁶ STAR -T cells/kg, employing a 3+3 escalation principle for dose titration. The primary objective of this study is to evaluate the safety of YTS109 cells therapy in treating recurrent/refractory autoimmune diseases, while the secondary objectives are to assess the efficacy of YTS109 cells as well as their pharmacokinetic and pharmacodynamic characteristics. The primary endpoint is observations of types, severity, and frequency of adverse events (AEs) and efficacy assessment. This single-arm, open-label trial will enroll patients across The First Affiliated Hospital of Anhui Medical University.

ELIGIBILITY:
Inclusion Criteria:

- Subjects must meet both the following common inclusion criteria and disease-specific inclusion criteria simultaneously to be eligible for participation in this study:

Common inclusion criteria:

1. Age ranges from 18 to 65 years old (including threshold), regardless of gender.
2. Essential Organ Function Criteria:

<!-- -->

1. Bone marrow: Neutrophils ≥1×10^9/L (within 2 weeks, excluding granulocyte colony-stimulating factor use); Hemoglobin ≥60 g/L.
2. Liver: ALT/AST ≤3×ULN (disease-related elevations permitted). TBIL≤1.5×ULN (disease-related elevations permitted).
3. Renal: CrCl≥30mL/min (Cockcroft-Gault formula, excluding acute declines).
4. Coagulation: INR/PT ≤1.5×ULN.
5. Cardiovascular: Hemodynamic stability. 3. Fertile females or males with partners of childbearing age must use medically approved contraception or abstain during and ≥12 months post- treatment. Negative serum HCG test (within 7 days pre-enrollment) for fertile females; non-lactating.

4. Voluntary participation with signed informed consent and compliance.

Specific inclusion criteria:

Relapsing and refractory systemic lupus erythematosus:

1. Meeting the 2019 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria for systemic lupus erythematosus (SLE); 2. Meeting the criteria for refractory lupus nephritis (LN) or SLE-associated immune thrombocytopenia (SLE-ITP), defined as follows:

1. Refractory Lupus Nephritis:

   ①Failure to achieve remission following treatment regimens comprising glucocorticoids and at least two immunosuppressive agents (including cyclophosphamide [CTX], tacrolimus, mycophenolate mofetil [MMF], and cyclosporine) and/or biologic agents (including rituximab, belimumab, telitacicept, etc.).
   * Urine protein-to-creatinine ratio (UPCR) ≥1.0 g/g or 24-hour urine protein excretion >1.0 g at screening.

     * Renal pathology must be performed within 6 months prior to the screening visit or during the screening period, demonstrating proliferative lupus nephritis (Class III or IV, with or without Class V) according to the 2003 International Society of Nephrology/Renal Pathology Society (ISN/RPS) criteria, with ≤50% glomerular sclerosis noted in the pathology report.
2. Refractory SLE-Associated Immune Thrombocytopenia:

   * Failure to achieve partial remission after at least one course of methylprednisolone pulse therapy (0.5-1 g × 3-5 days) or high-dose glucocorticoids (equivalent to 1 mg/kg/day of prednisone) combined with one or more immunosuppressive agents (including biologic agents) for at least 3 months, or inability to maintain therapeutic efficacy during glucocorticoid tapering. Platelet count <50 × 10⁹/L on at least two consecutive complete blood count tests prior to enrollment. Exclusion of thrombocytopenia due to non-SLE causes, such as infection, bone marrow suppression, or hypersplenism.

Relapsing and refractory Sjögren's syndrome:

1. Meeting the 2002 American-European Consensus Group (AECG) criteria or the 2016 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) classification criteria for primary Sjögren's syndrome; 2. Having a disease activity score of EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) ≥ 6; 3. Testing positive for anti-SSA/Ro antibodies; 4. Definition of relapsing and refractory condition: Persistence of disease activity or recurrence of disease activity after remission, despite undergoing conventional treatment for more than six months. Definition of conventional treatment: Administration of glucocorticoids in combination with any of the following immunosuppressive agents or biological agents: cyclophosphamide, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, as well as biological agents including rituximab, belimumab, telitacicept, etc.

Relapsing and refractory Sjogren's Syndrome:

1. Meeting the 2013 American College of Rheumatology (ACR) classification criteria for systemic sclerosis;
2. Testing positive for systemic sclerosis-related antibodies;
3. Presenting with diffuse cutaneous sclerosis or active interstitial lung disease (as indicated by ground-glass opacities on high-resolution computed tomography, HRCT);
4. Definition of relapsing and refractory condition: Persistence of disease activity or recurrence of disease activity after remission, despite undergoing conventional treatment for more than six months. Definition of conventional treatment: Administration of glucocorticoids and cyclophosphamide, in combination with any one or more of the following immunomodulatory agents: antimalarial drugs, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, as well as biological agents including rituximab, belimumab, telitacicept, etc.;
5. Definition of progressive condition: Demonstrating rapid skin progression (an increase in modified Rodnan skin score, mRSS, of >25%) or pulmonary disease progression (a 10% decrease in forced vital capacity, FVC, or a >5% decrease in FVC accompanied by a 15% decrease in diffusion capacity for carbon monoxide, DLCO).

Note: Meeting either criterion 4 or 5 is sufficient.

Relapsing and refractory Inflammatory Myopathy:

1. Meeting the 2017 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria for inflammatory myopathies (including dermatomyositis, DM; polymyositis, PM; antisynthetase syndrome, ASS; and necrotizing myopathy, NM); 2. Testing positive for myositis-specific antibodies; 3. For patients with muscle involvement, having a Manual Muscle Testing-8 (MMT-8) score below 142 and at least two abnormal findings among the following five core measures (Physician's Global Assessment, PhGA; Patient's Global Assessment, PtGA, or extra-muscular disease activity score ≥ 2 points; Health Assessment Questionnaire, HAQ, total score ≥ 0.25; muscle enzyme levels 1.5 times the upper limit of normal range); or having an MMT-8 score ≥ 142 but presenting with active interstitial lung disease (as indicated by ground-glass opacities on high-resolution computed tomography, HRCT); 4. Definition of relapsing and refractory condition: Persistence of disease activity or recurrence of disease activity after remission, despite undergoing conventional treatment for more than six months. Definition of conventional treatment: Administration of glucocorticoids and cyclophosphamide, in combination with any one or more of the following immunomodulatory agents: antimalarial drugs, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, as well as biological agents including rituximab, belimumab, telitacicept, etc.; 5. Definition of progressive condition: Demonstrating worsening myositis or rapidly progressive interstitial pneumonia.

Note: Meeting either criterion 4 or 5 is sufficient.

Relapsing and refractory Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis:

1. Meeting the 2022 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) diagnostic criteria for ANCA-associated vasculitis, including microscopic polyangiitis, granulomatosis with polyangiitis, and eosinophilic granulomatosis with polyangiitis.

2. Testing positive for ANCA-related antibodies (either MPO-ANCA or PR3-ANCA positive).

3. A Birmingham Vasculitis Activity Score (BVAS) of ≥15 points (out of a total of 63 points), indicating active vasculitis.

4. Definition of relapsing/refractory condition: Persistence of disease activity or recurrence of disease activity after remission, despite undergoing conventional treatment for more than six months. Definition of conventional treatment: Administration of glucocorticoids and cyclophosphamide, in combination with any one or more of the following immunomodulatory agents: antimalarial drugs, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, as well as biological agents including rituximab, belimumab, telitacicept, etc.

Relapsing and refractory Antiphospholipid Syndrome:

1. Meeting the 2006 Sydney-revised diagnostic criteria for primary antiphospholipid syndrome; 2. Testing positive for antiphospholipid antibodies at moderate to high titers (IgG/IgM antibodies against lupus anticoagulant, LA; beta-2 glycoprotein I, B2GP1; or anticardiolipin, acL, detected positive on more than two occasions within a 12-week period); 3. Definition of relapsing/refractory condition: Recurrence of thrombosis despite standard treatment with warfarin anticoagulation or alternative vitamin K antagonist (i.e., maintaining the required international normalized ratio, INR, for therapeutic management) or standard therapeutic doses of low molecular weight heparin (LMWH), in addition to previous treatment with corticosteroids and cyclophosphamide; 4. For catastrophic antiphospholipid syndrome, the following four criteria must be met: (1) involvement of three or more organs, systems, and/or tissues; (2) onset of symptoms within one week; (3) histological confirmation of small vessel occlusion in at least one organ or tissue; (4) presence of aPL (antiphospholipid antibodies).

Note: Meeting either criterion 3 or 4 is sufficient.

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria will not be admitted to the study:

  1. Individuals with a severe history of drug allergies or those with an allergic constitution;
  2. Individuals with existing or suspected uncontrolled or treatable fungal, bacterial, viral, or other infections;
  3. Subjects with central nervous system diseases (excluding those with a history of epilepsy, psychiatric disorders, organic brain disease syndromes, cerebrovascular accidents, encephalitis, or central nervous system vasculitis resulting from the underlying disease);
  4. Subjects whose cardiac function cannot tolerate the study interventions;
  5. Subjects with congenital immunoglobulin deficiencies;
  6. Subjects with a history of malignant tumors within the past five years;
  7. Subjects with end-stage renal failure;
  8. Subjects who are positive for hepatitis B surface antigen (HBsAg) and hepatitis B core antibody (HBcAb) with peripheral blood HBV DNA titers exceeding the upper limit of detection; subjects who are positive for hepatitis C virus (HCV) antibody and peripheral blood HCV RNA; subjects who are positive for human immunodeficiency virus (HIV) antibody; and subjects who are positive for syphilis testing;
  9. History of symptomatic deep vein thrombosis or pulmonary embolism within the 6 months prior to screening;
  10. Subjects with psychiatric disorders or severe cognitive dysfunction;
  11. Subjects who have participated in other clinical trials within the past three months prior to enrollment;
  12. Subjects who have received immunosuppressive agents with therapeutic effects on the disease within five half-lives prior to enrollment or biological agents within four weeks prior to enrollment;
  13. Pregnant women or women planning to become pregnant;
  14. Subjects whom the investigator believes have other reasons that preclude their inclusion in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-11-13 (Estimated); Primary Completion 2026-11-13 (Estimated); Study Completion 2027-11-13 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | The efficacy endpoint evaluation for 2, 4, 8, 12 weeks, AEs observation will be follow-up for 24 weeks. The observation period is extended to 52 weeks.
  1. Types, severity, and frequency of adverse events (AEs);
  2. Incidence of dose-limiting toxicity (DLT).

SECONDARY OUTCOMES:
Efficacy Evaluation in relapsed/refractory autoimmune diseases | 2, 4, 8, 12 weeks, and the observation will continue until 24 to 52 weeks post-treatment.
  The proportion of subjects achieving complete response (CR), partial response (PR), or other responses at week 12.
Maximum Plasma Concentration of YTS109 (Cmax) | The detections will be conducted on day0, 4, 7, 10, and weeks 2, 3, 4, 8, 12. Then, observation will continue until 12 to 24 weeks post-treatment.
  To evaluate the metabolic characteristics of YTS109
Area Under the Plasma Concentration-Time Curve (AUC) of YTS109 | The detections will be conducted on day0, 4, 7, 10, and weeks 2, 3, 4, 8, 12. Then, observation will continue until 12 to 24 weeks post-treatment.
  To evaluate the metabolic characteristics of YTS109
Time to Reach Maximum Plasma Concentration (Tmax) of YTS109 | The detections will be conducted on day0, 4, 7, 10, and weeks 2, 3, 4, 8, 12. Then, observation will continue until 12 to 24 weeks post-treatment.
  To evaluate the metabolic characteristics of YTS109
Cytokines Concentration Level Change | The detections will be conducted on day0, 4, 7, 10, and weeks 2, 3, 4, 8, 12. Then, observation will continue until 24 to 52 weeks post-treatment.
  Evaluate the Pharmacodynamic (PD) effects of YTS109 cells
The reconstitution of B cell in peripheral blood | The detections will be conducted on day0, 4, 7, 10, and weeks 2, 3, 4, 8, 12. Then, observation will continue until 24 to 52 weeks post-treatment.
  Changes in B cells quantification and phenotypic in peripheral blood